CLINICAL TRIAL: NCT01236144
Title: An NCRI Acute Myeloid Leukaemia Working Group Pilot Trial Under the Auspices of the Cardiff Experimental Cancer Medicine Centre to Establish the Feasibility of Combining Either the Tyrosine Kinase Inhibitor AC220,CXCR4 Inhibitor Plerixafor or HSP90 Inhibitor Ganetespib With Chemotherapy in Older Patients With Acute Myeloid Leukaemia and High Risk Myelodysplastic Syndrome.
Brief Title: A Trial to Establish the Feasibility of Combining Either the Tyrosine Kinase Inhibitor AC220,CXCR4 Inhibitor Plerixafor or HSP90 Inhibitor Ganetespib With Chemotherapy in Older Patients With Acute Myeloid Leukaemia and High Risk Myelodysplastic Syndrome.
Acronym: AML18 Pilot
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cardiff University (Other)
Collaborators: Leukaemia & Lymphoma Research Group (Unknown); Experimental Cancer Medicine Centres (Other)
Responsible Party: Principal Investigator, Alan K Burnett, Chief Investigator, Cardiff University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPON 845-10; 2010-021444-18 (EudraCT Number); 10/MRE09/27 (Other: Research Ethics Committee for Wales)
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Acute Myeloid Leukaemia; High Risk Myelodysplastic Syndrome
Keywords: Myeloid; Leukaemia; Acute; Myelodysplastic; Pilot; Cardiff; Haematology; Burnett; AC220; Plerixafor; Ganetespib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — plerixafor; STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AC220 Intervention (Experimental)
  Interventions: Drug: AC220
- Plerixafor Intervention (Experimental)
  Interventions: Drug: Plerixafor
- Ganetespib (Experimental)
  Interventions: Drug: Ganetespib

INTERVENTIONS:
Drug: Plerixafor — Fixed dose of Plerixafor (240mcg/kg) given by subcutaneous injection on each day of chemotherapy for up to 3 courses (depending on cohort). The three chemotherapy courses will be Daunorubicin/Clofarabine for courses 1&2 and Daunorubicin/Ara-C for course 3. Each course will last 5 days, and Plerixafor will be given for 5 days.
  Other Names: Mozobil
  Arms: Plerixafor Intervention
Drug: AC220 — Each cohort of patients will receive three courses of chemotherapy approximately 4 to 5 weeks apart which will comprise of Daunorubicin/Ara-C/Etoposide in Courses 1&2 and Daunorubicin/Ara-C in Course 3. Two days after the last day of each chemotherapy course, patients will receive AC220 orally for 7, 14 or 21 (depending on cohort) consecutive days. Depending on which cohort the patient enters, they will receive either 60mg, 90mg or 135mg of AC220 daily, with a provision to assess 40mg if necessary.
  Arms: AC220 Intervention
Drug: Ganetespib — Patients will receive 3 treatments of ganetespib on days 1, 8 and 15 of each course where day 1 is the first day of the chemotherapy. The chemotherapy will be DAE/DAE/DA. Three courses of chemotherapy will be given each of which will be associated with 3 administrations of ganetespib.
  Arms: Ganetespib

SUMMARY:
The AML18 Pilot Trial will evaluate the feasibility of three interventions that are planned to be included in the forthcoming NCRI AML18 Trial. One intervention will be to evaluate combining the Tyrosine Kinase Inhibitor AC220 with three courses of standard DAE (Daunorubicin, Ara-C, Etoposide). AC220 will be given following each treatment course, daily by mouth for 7, 14 or 21 days. AC220 will be evaluated at 3 dose levels of 60, 90 and 135 mg flat dose. A 4th dose level of 40 mg will be introduced should patients not respond well to 60 mg. The second intervention to be tested is the combination of the CXCR4 inhibitor Plerixafor with up to three courses of the chemotherapy combination of DClo (Daunorubicin, Clofarabine). Patients/investigators will be able to choose which intervention to enter. Depending on recruitment requirements, only one intervention might be available at any one time. The third intervention Patients will receive 3 treatments of 100 mg of ganetespib on days 1, 8 and 15 of each course where day 1 is the first day of the chemotherapy. The chemotherapy will be DAE/DAE/DA. Three courses of chemotherapy will be given each of which will be associated with 3 administrations of ganetespib.

DETAILED DESCRIPTION:
The AML18 Pilot Trial is available to any patient who has primary or secondary AML as defined by the WHO Classification (Appendix A) (excluding Acute Promyelocytic Leukaemia), or high risk Myelodysplastic Syndrome (i.e. > 10% marrow blasts) who is not considered suitable for the current NCRI trial for younger patients (MRC AML 17). This trial has the primary aim of assessing the feasibility of three treatments that are planned for the forthcoming NCRI AML18 Trial. The first is the feasibility of adding AC220, given sequentially initially for 7 days, to three courses of standard chemotherapy. AC220 will be assessed at up to three daily dose levels: - 60mg/day, 90mg/day, 135 mg/day and also, if required, at 40mg/day. The protocol will also assess in a separate study cohort the feasibility of combining the CXCR4 inhibitor, Plerixafor, at a fixed dose in combination with up to three courses of chemotherapy. The third intervention patients will receive 3 treatments of ganetespib on days 1, 8 and 15 of each course where day 1 is the first day of the chemotherapy. The chemotherapy will be DAE/DAE/DA. Three courses of chemotherapy will be given each of which will be associated with 3 administrations of ganetespib.

THERAPEUTIC INTERVENTIONS

Therapeutic Interventions for AC220 Assessment:

Patients will enter one of 3 dose level cohorts either 60mg/day, 90mg/day or 135mg/day with the provision to assess 40mg/day if required. Each cohort will receive three courses of chemotherapy approximately 4 to 5 weeks apart, which will comprise DAE ( Daunorubicin, Ara-C, Etoposide) over 10 days (Course 1) , DAE over 8 days (Course 2) and DA (Daunorubicin, Ara-C) over 5 days (Course 3). Two days after the last day of chemotherapy patients will receive the AC220 orally, daily for 7 consecutive days. Formal safety and pharmaco-kinetic assessments will be undertaken on day 1, 7 and 14 of each course of AC220, and interim toxicities will also be required to be reported. Sufficient patients must enter each AC220 dose level cohort to ensure that at least 3 patients are evaluable for all three courses. Cohort 2 (i.e.60mg/day for 14 days) can open to recruitment after a minimum of 3 evaluable patients have completed course 1. Cohort 3 (40mg/day dose level for either 7/14 days) will be undertaken if cohort 1 or 2 are unsuccessful i.e. fail to satisfy the safety criteria.

It is anticipated that the 'study dose' will be established from the experience of cohorts 1 to 5. Cohort 6 ('study dose') will receive AC220 for 21 days after each chemotherapy course. In this cohort there must be a minimum of a 10 days break between the end of the AC220 course and the start of the subsequent chemotherapy course.

Therapeutic Interventions for Plerixafor Assessment:

The aim is to assess the feasibility of combining a fixed dose (240mcg/kg) of Plerixafor given on each day of chemotherapy for up to 3 courses, and if so to combine this with G-CSF in courses 2 and 3. The three chemotherapy courses will be Daunorubicin/Clofarabine (DClo) for courses 1 & 2 and Daunorubicin/Ara-C (DA) for course 3. Each course will last 5 days and Plerixafor will be given for 5 days.

Cohort 1 will receive three courses of chemotherapy with Plerixafor in course 1 only. Cohort 2 will receive three courses with Plerixafor in course 1 and 2. Cohort 3 will receive chemotherapy with Plerixafor in all three courses. Cohort 4 will be the same as cohort 3 but they will also receive G-CSF in course 2 and 3.

Therapeutic Interventions for Ganetespib Assessment:

There will be one feasibility cohort of 10 evaluable patients who require to be evaluable after 30 days after the first course, where day 1 is the first day of chemotherapy. Patients will receive 3 treatments of ganetespib on days 1, 8 and 15 of each course where day 1 is the first day of the chemotherapy. The chemotherapy will be DAE/DAE/DA. Three courses of chemotherapy will be given each of which will be associated with 3 administrations of ganetespib.

ELIGIBILITY:
Inclusion Criteria:

* They have one of the forms of acute myeloid leukaemia, except Acute Promyelocytic Leukaemia or CML in blast crisis as defined by the WHO Classification (Appendix A) - this can be any type of de novo or secondary AML - or high risk Myelodysplastic Syndrome, defined as greater than 10% marrow blasts (RAEB-2).
* Serum creatinine ≤ 1.5 × ULN (upper limit of normal)
* White cell count of <30 x 109/L at diagnosis (for Plerixafor option only). If WCC is >30 x 109/l patients in the Plerixafor pilot should have the WCC reduced to <30 x 109/L using Hydroxycarbamide to avoid the risk of hyperleucocytosis
* Serum potassium, magnesium, and calcium levels should be at least within institutional normal limits, and every effort should be made to keep potassium at institutional normal limits, and every effort should be made to keep potassium concentrations above 4.0 mEq/dL, and serum calcium at normal concentration.
* Total serum bilirubin ≤ 1.5 × ULN (upper limit of normal) and serum aspartate transaminase (AST) and/or alanine transaminase (ALT) ≤ 2.5 × ULN
* Sexually mature males must agree to use an adequate and medically accepted method of contraception throughout the study if their sexual partners are women of child bearing potential (WOCBP).
* Over 60 years of age
* Provided written informed consent

Exclusion Criteria:

* They have previously received cytotoxic chemotherapy for AML. [Hydroxycarbamide, or similar low-dose therapy, to control the white count prior to initiation of intensive therapy is not an exclusion].
* They are in blast transformation of chronic myeloid leukaemia (CML).
* They have a concurrent active malignancy excluding basal cell carcinoma.
* They are pregnant or lactating.
* They have Acute Promyelocytic Leukaemia
* Known infection with human immunodeficiency virus (HIV)

Patients are not eligible for the AC220 option if they have:

* Uncontrolled or significant cardiovascular disease, including :
* A myocardial infarction within 12 months
* Uncontrolled angina within 6 months
* Current or history of congestive heart failure New York Heart Association (NYHA) class 3 or 4, unless an echocardiogram (ECHO) or Multiple Gated Acquisition Scan (MUGA) performed either within 1 month prior to study screening or during screening results in a left ventricular ejection fraction (LVEF) that is ≥ 45% (or institutional lower limit of normal value).
* Diagnosed or suspected congenital long QT syndrome. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes [TdP]); any history of arrhythmia will be discussed with the Sponsor's Medical Monitor prior to patient's entry into the study.
* Prolonged QTcF interval on pre-entry ECG (≥450 ms) - this will be the average of 3 readings within a 2 hour period.
* Any history of second or third degree heart block (may be eligible if the patient currently has a pacemaker).
* Heart rate < 50/minute on pre-entry ECG
* Uncontrolled hypertension
* Obligate need for a cardiac pacemaker
* Complete left bundle branch block
* Atrial fibrillation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Response (CR, CRi, PR) achievement, and reasons for failure | Duration of treatment
Mortality | At 30 days and 8 weeks
Toxicity (haematological and non-haematological) | Duration of trial treatment
Survival | At 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alan K Burnett, Study Chair — Cardiff University; Nigel H Russell, Study Chair — Nottingham University
Locations (13):
- United Kingdom (13):
  - Aberdeen Royal Infirmary, Aberdeen
  - Belfast City Hospital, Belfast
  - Birmingham Heartlands Hospital, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Castle Hill Hospital, Hull
  - St James's University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - St Bartholomew's Hospital, London
  - Christie Hospital, Manchester
  - Manchester Royal Infirmary, Manchester
  - Freeman Hospital, Newcastle
  - Nottingham University Hospital, Nottingham